CLINICAL TRIAL: NCT02035995
Title: EVALUATION OF THE MACULAR, PERIPAPILLARY NERVE FIBER LAYER AND CHOROID THICKNESS CHANGES IN THE GESTATIONAL DIABETES MELLITUS, HEALTHY PREGNANT AND WOMEN VOLUNTEERS.
Status: Completed | Type: Observational
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gökhan Açmaz, MD, Kayseri Education and Research Hospital
Other Study IDs: GokhanAcmaz
Record Dates: First submitted 2014-01-11; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Retinal Evaluation in Patients With GDM.
Keywords: gestational diabetes mellitus; optical coherence tomography; pregnancy; retinal nerve fiber layer.
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: None Retained — no biospecimens are to be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy volunteers: This group consisted of age matched non-pregnant healthy volunteers
  Interventions: Other: Pregnant volunteers with GDM
- Healthy pregnant volunteers: This group consisted of age matched healthy pregnant volunteers
  Interventions: Other: Pregnant volunteers with GDM

INTERVENTIONS:
Other: Pregnant volunteers with GDM

SUMMARY:
Gestational diabetes mellitus (GDM) is a risk factor for the development of type II diabetes and it is responsible for the morbidity of both mother and child. The aim of this study was to determine retinal findings of gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
We have three groups; the first group consisted of pregnant volunteers with GDM. The second group consisted of healthy pregnant participants. The third group consisted of healthy, non-pregnant women at the reproductive age. Macular, choroid and retinal nerve fiber layer (RNFL) thicknesses were evaluated in patients with GDM and comparisons were made among GDM, healthy pregnant and healthy non-pregnant subjects for these parameters by using optic cohorence tomography.

ELIGIBILITY:
Inclusion Criteria:

Singleton pregnancies Pregnancies between 26-28 weeks of gestation Gestational Diabetes

Exclusion Criteria:

* ocular surgery ocular trauma glaucoma cystoid macular edema macular degeneration optic atrophy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Retinal evaluation | 6 weeks
  The aim of this study was to determine retinal findings of gestational diabetes mellitus (GDM).

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri Education and Research Hospital, Kayseri, Turkey (Türkiye)